CLINICAL TRIAL: NCT03347526
Title: A Novel Approach to Infantile Spasms: Combined Cosyntropin Injectable Suspension, 1 mg/mL and Vigabatrin Induction Therapy
Brief Title: A Novel Approach to Infantile Spasms
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: Study on enrollment hold as a precaution per the pharmaceutical company.
Sponsor: University of Colorado, Denver (Other)
Collaborators: Pediatric Epilepsy Research Foundation (Unknown); West Therapuetics, Inc (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-0222
Record Dates: First submitted 2017-11-15; First posted 2017-11-20 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Infantile Spasm
Keywords: Vigabatrin; Cosyntropin
MeSH Terms: conditions — Spasms, Infantile | interventions — Vigabatrin

STUDY DESIGN:
Masking Description: Blinded outcome measure
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cosyntropin Injectable Suspension, 1mg/mL + vigabatrin (Experimental)
  Interventions: Drug: Cosyntropin Injectable Suspension 1 MG/ML + vigabatrin
- Cosyntropin Injectable Suspension, 1 mg/mL (Experimental)
  Interventions: Drug: Cosyntropin Injectable Suspension, 1 mg/mL
- Vigabatrin (Active Comparator)
  Interventions: Drug: Vigabatrin

INTERVENTIONS:
Drug: Cosyntropin Injectable Suspension, 1 mg/mL — Injectable
  Arms: Cosyntropin Injectable Suspension, 1 mg/mL
Drug: Cosyntropin Injectable Suspension 1 MG/ML + vigabatrin — Injectable + oral solution
  Arms: Cosyntropin Injectable Suspension, 1mg/mL + vigabatrin
Drug: Vigabatrin — oral
  Arms: Vigabatrin

SUMMARY:
This study proposes to assess the efficacy of Cosyntropin Injectable Suspension, 1 mg/mL compared to vigabatrin. Additionally, this study proposes to determine efficacy of combination therapy of Cosyntropin Injectable Suspension, 1 mg/mL and vigabatrin to monotherapy Cosyntropin Injectable Suspension, 1mg/mL in children with new onset infantile spasms (IS).

DETAILED DESCRIPTION:
This is a prospective randomized trial comparing 3 treatment arms:

1. Cosyntropin Injectable Suspension, 1 mg/mL
2. Vigabatrin
3. Combination of both these therapies, Cosyntropin Injectable Suspension, 1 mg/mL and vigabatrin for treatment of new onset infantile spasms. Outcome measures include resolution of clinical spasms, improvement of hypsarrhythmia as well as longer term outcomes of development and subsequent seizures.

The data is expected to demonstrate greater efficacy with Cosyntropin Injectable Suspension, 1 mg/mL than vigabatrin for the treatment of IS.

ELIGIBILITY:
Inclusion Criteria:

* New onset infantile spasms
* Age > 2 months
* Age< 2 years
* Hypsarrhythmia on video-EEG
* Normal renal function

Exclusion Criteria:

* Prior treatment given for infantile spasms
* Diagnosis of Ohtahara syndrome or Early Myoclonic Epilepsy
* Absence of hypsarrhythmia
* Inability for the parent or caregiver to provide consent
* Inability for the parent or caregiver to complete seizure diary
* Diagnosis of:

  * scleroderma,
  * osteoporosis,
  * recent systemic fungal infections,
  * ocular herpes simplex,
  * recent surgery,
  * history of or the presence of a peptic ulcer,
  * congestive heart failure,
  * uncontrolled hypertension

Ages: 2 Months to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 394 (Estimated)
Dates: Start 2018-04-19 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
A comparison of Cosyntropin Injectable Suspension and Vigabatrin on the proportion of subjects who become spasm-free as defined by a) and b). | 2 weeks
  a) Resolution of hypsarrhythmia via video electroencephalogram (EEG), and b) Resolution of clinical spasms via video EEG.

SECONDARY OUTCOMES:
A comparison of combination therapy and Cosyntropin Injectable Suspension alone (monotherapy) on the proportion of subjects who become spasm-free as defined by a) and b) | Day 14-42
  a) Resolution of clinical spasms for 48 hours at 2 weeks sustained until day 42, and b) Resolution of hypsarrhythmia via video EEG at 2 weeks.
A comparison between combination therapy and Cosyntropin Injectable Suspension alone (monotherapy) on the proportion of subjects who become seizure free at 6 months. | 6 months
  Difference in proportion of subjects who are seizure free between 5 and 6 months after treatment.
Comparison between combination therapy and Cosyntropin Injectable Suspension alone (monotherapy). | 18 months chronological age
  A comparison between combination therapy and Cosyntropin Injectable Suspension alone (monotherapy) on developmental scores as measured by the Adaptive Behavior Assessment System (ABAS III) at 18 months chronological age.
Comparison between combination therapy and Cosyntropin Injectable Suspension alone (monotherapy). | 18 months chronological age
  A comparison between combination therapy and Cosyntropin Injectable Suspension alone (monotherapy) on developmental scores as measured by the Vineland II at 18 months chronological age.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly G. Knupp, MD, Principal Investigator — University of Colorado, Denver
Locations (14):
- United States (14):
  - Children's Hospital Los Angeles, Los Angeles, California
  - UCSF Medical Center, San Francisco, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta at Scottish Rite, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - C.S. Mott Children's Hospital, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Columbia University Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Atrium Health, Charlotte, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - Cook Children's Medical Center, Fort Worth, Texas

IPD SHARING:
Plan to Share IPD: Undecided